CLINICAL TRIAL: NCT04649918
Title: Short and Medium-term Effects of Pulmonary Rehabilitation in Mild to Critical Post-acute COVID-19 - an Observational Trial
Brief Title: Short and Medium-term Effects of Pulmonary Rehabilitation in Mild to Critical Post-acute COVID-19
Acronym: STEPCO
Status: Completed | Type: Observational
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Professor, Schön Klinik Berchtesgadener Land
Other Study IDs: COVID-Rehab
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Covid19; SARS-CoV Infection; Pulmonary Rehabilitation; Quality of Life
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mild to moderate COVID 19: patients post-acute mild to moderate COVID 19
  Interventions: Other: pulmonary rehabilitation
- severe to critical COVID 19: patients post-acute severe to critical COVID 19
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — COVID 19 patients perform a standardized 3-week inpatient pulmonary rehabilitation program

SUMMARY:
As a direct consequence of the COVID-19 pandemic, it is assumed that the number of patients with COVID-19-related disabilities will increase significantly. Patients with mild, severe, and critical forms of the disease show long-term sequelae in different systems (respiratory, muscular, psychological, cognitive etc.).

Persistent dyspnea is a frequently described symptom after the acute phase of the disease. Coupled with reduced oxygen saturation, an increased risk of developing lung fibrosis has been observed. Specialized rehabilitation medicine (e.g. pulmonary rehabilitation) might counteract these long-term consequences and therefore seems to be a promising approach to treat long-term COVID-19 consequences.

Further, there is scarce evidence about COVID-19 specific rehabilitation contents. It was suggested to use treatment regimes in analogy to patients with idiopathic pulmonary fibrosis.

There is evidence that pulmonary rehabilitation improves physical performance, quality of life and reduces anxiety and depression symptoms in patients with idiopathic pulmonary fibrosis and other chronic respiratory diseases.

Since impairments related to idiopathic pulmonary fibrosis also play an important role in COVID-19, the aim of this study is to evaluate the short and medium-term effects of a standardized 3-week pulmonary rehabilitation program. The results will be analyzed within the two cohorts (mild/moderate and severe/critical COVID 19) as well as between the two cohorts for the primary outcome. Furthermore, the effects of pulmonary rehabilitation will be compared with a retrospective cohort of idiopathic pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Post-acute phase COVID-19 patients with mild, moderate, severe or critical course
* written informed consent

Exclusion Criteria:

* patients who are unable to walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred for an inpatient pulmonary rehabilitation program at the reference center will be recruited
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | Day 1 and day 21 of pulmonary rehabilitation
  measure in meter

SECONDARY OUTCOMES:
change in endurance shuttle walk distance | Day 1 and day 21 of pulmonary rehabilitation
  measure provided in seconds
Change in Diffusion capacity of the lungs for Carbon monoxide | Day 1 and day 21 of pulmonary rehabilitation
  measure provided in % predicted
Change in Forced Vital Capacity | Day 1 and day 21 of pulmonary rehabilitation
  measure provided in % predicted
Change in total lung capacity | Day 1 and day 21 of pulmonary rehabilitation
  measure provided in % predicted
change in Montreal cognitive assessment test | Day 1 and day 21 of pulmonary rehabilitation
  score ranges from 0 to 30 with lower score indicating higher cognitive impairment
change in short-form 36 question health survey | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  score ranges from 0 to 100 with higher scores indicating better Quality of life
change in Patient-Reported Outcomes Measurement Information System - 29 (PROMIS-29) | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  A questionnaire designed to measure self-reported physical, mental and social health and wellbeing. Higher scores represent worse symptomatology in relation to the mean value of 50 points with a standard deviation of 10 points.
Change in the scale of general anxiety disorder - 7 questionnaire (GAD-7) | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  score ranges from 0 to 21 with higher scores indicating more severe anxiety
Change in the scale of the patient health questionnaire - Depression (PHQ-D) | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  score ranges from 0 to 27 with higher scores indicating more severe depression
Change in prevalence of COVID-19 related dyspnea | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  patients will be asked if they still perceive COVID-19 related dyspnea: answer possibilities yes or no
Change in prevalence of COVID-19 related cough | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  patients will be asked if they still perceive COVID-19 related cough: answer possibilities yes or no
Change in prevalence of COVID-19 related cognitive impairment | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  patients will be asked if they still perceive COVID-19 related cognitive impairment: answer possibilities yes or no
Change in prevalence of COVID-19 related loss of appetite | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  patients will be asked if they still perceive COVID-19 related loss of appetite: answer possibilities yes or no
Change in general perceived well-being | Day 1 and day 21 of pulmonary rehabilitation and day 90 following pulmonary rehabilitation
  scale from 1 (worst) to 10 (best)
change in D-Dimer level | Day 1 and day 21 of pulmonary rehabilitation
  in mg/l
change in c-reactive protein level | Day 1 and day 21 of pulmonary rehabilitation
  in mg/l
change in leukocytes level | Day 1 and day 21 of pulmonary rehabilitation
  in g/l
change in hemoglobin level | Day 1 and day 21 of pulmonary rehabilitation
  in g/dl
change in troponin level | Day 1 and day 21 of pulmonary rehabilitation
  in pg/ml
change in pro-brain natriuretic peptide level | Day 1 and day 21 of pulmonary rehabilitation
  in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Koczulla, MD, Principal Investigator — Philipps University Marburg
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided